CLINICAL TRIAL: NCT00801606
Title: Micronutrient Supplementation in Conjunction With Standard Anti-Tuberculosis Therapy in Paediatric (6 Months-15 Years) New Pulmonary Tuberculosis Patients
Brief Title: Micronutrient Supplementation in in Paediatric Pulmonary Tuberculosis
Acronym: ICTBSG
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: All India Institute of Medical Sciences (Other)
Collaborators: University of Bergen (Other)
Responsible Party: Principal Investigator, SK Kabra, Dr, All India Institute of Medical Sciences
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ICTBSG
Record Dates: First submitted 2008-12-02; First posted 2008-12-03 (Estimated); Last update posted 2016-02-10 (Estimated); Status verified 2016-02

CONDITIONS: Tuberculosis
Keywords: Micronutrient; Childhood Tuberculosis
MeSH Terms: conditions — Tuberculosis | interventions — Zinc; Drug Evaluation; Micronutrients

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Study drug containing zinc alone (Experimental): Zinc 20 mg daily
  Interventions: Drug: Zinc
- Study drug Micronutrient without zinc (Experimental): micronutrients (vitamin A, thiamine, riboflavin, vitamins B-6 and B-12, folic acid, niacin, vitamins C, E, and D, selenium, and copper) without zinc.
  Interventions: Drug: Micronutrient without zinc
- Study drug Micronutrient with zinc (Experimental): micronutrients in combination with zinc (vitamin A, thiamine, riboflavin, vitamin B-6 and B-12, folic acid, niacin, vitamins C, E, and D, selenium, copper, and 20 mg elemental zinc).
  Interventions: Drug: Micronutrient with zinc
- Placebo (Placebo Comparator): Placebo only
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Zinc — Zinc 20 mg/day
  Other Names: study drug
  Arms: Study drug containing zinc alone
Drug: Micronutrient without zinc — Multimineral 2 RDA
  Other Names: study drug
  Arms: Study drug Micronutrient without zinc
Drug: Micronutrient with zinc — Multimineral 2 RDA and zinc 20 mg per day
  Other Names: study drug
  Arms: Study drug Micronutrient with zinc
Drug: Placebo — Placebo
  Other Names: study drug
  Arms: Placebo

SUMMARY:
A recent trial in adults has demonstrated that zinc (Zn) and other Multiminerals (MN) combined, but neither of them alone, significantly increased weight gain during Tuberculosis (TB) treatment. There was a substantially larger beneficial effect on survival amongst those who received the combination of Zn and MN compared with those who received either Zn alone or MN alone. These exciting preliminary findings require further confirmation, as the data on mortality reduction was based on a post-hoc subgroup-analysis. Effects of MN and Zn supplementation has not been assessed in children with TB. Studies are urgently needed to evaluate the therapeutic potential of nutritional interventions on treatment outcome in children with TB. Simple and inexpensive nutritional interventions may substantially impact TB-related child morbidity and mortality in high-burden settings. The investigators thus, propose a randomized, double blind, controlled trial that will measure the effect of multi-vitamin/mineral supplementation on the efficacy of anti-TB treatment in newly diagnosed childhood pulmonary TB patients in Delhi.

DETAILED DESCRIPTION:
We plan to do a randomized controlled trial to study impact of multimineral supplement with antituberculosis drugs in freshly diagnosed pulmonary tuberculosis in children. Plan to enrol 400 children at two sites in Delhi. The diagnosis and treatment of pulmonary tuberculosis will be based on recommendations of Revised National Tuberculosis Control Program (RNTCP). The outcome will be measured in form of weight gain and improvement in x ray film of chest. The secondary outcome variables will be as follows:

1. Effect of micronutrient supplements at 2 and 6 months on anthropometric parameters by comparing means of anthropometric parameters in different groups.
2. Improvement in radiological findings at 2 months: Comparing the proportion of children showing clearance of X ray films at baseline and 6 months by two paediatricians independently using same protocol.
3. Resolution of symptoms at 2 and 6 months: By comparing proportion of patients having resolution of presenting symptoms (fever, cough, appetite improvement) as reported by parents
4. Proportion of children requiring extension of intensive phase of therapy: Comparing proportion of children in different groups requiring extension of intensive phase of therapy at 2 months due to the treating physician's decision.
5. Interferon gamma responses to M. tuberculosis antigens ESAT6 and CF10 by quantiferon assay at baseline, 2 months and 6 months of treatment
6. To study effect of zinc supplementation on ocular toxicity in children receiving ethambutol by VER
7. To document drug resistance (S, I, R, E) patterns among children with culture confirmed TB
8. To document genotypic strain diversity among children with culture confirmed TB, also associations between strain type and disease severity and/or drug resistance
9. To document the spectrum of mycobacterial species by culture in children clinically suspected of having pulmonary tuberculosis.

ELIGIBILITY:
Inclusion Criteria:

* New pulmonary (including pleural) tuberculosis with/without an extrapulmonary lesion in children age 6 months to 15 years

Exclusion Criteria:

* Weight for height < 70 % of NCHS median (reason: zinc as per guidelines is given as standard point of care to all severely malnourished children)
* Bilateral pedal oedema
* Known HIV + ve
* Place of residence outside Delhi (including physicians discretion)
* History of previous ATT treatment or INH prophylaxis for more than 48 hours prior to enrollment
* Signs of upper airway obstruction, or an arterial oxygen saturation less than 92% in room air
* Signs of renal, hepatic, or cvs disease
* Unable to attend follow up session for reading of Mantoux tests
* Documented intake of zinc continuously for > 2 weeks in the preceding 4 weeks at enrollment
* CNS, osteo-articular, pericardial, renal TB
* History of contact with a documented case of drug resistant TB

Ages: 6 Months to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 403 (Actual)
Dates: Start 2008-12; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Change in Z score for weight and improvement in X ray film | 6 months

SECONDARY OUTCOMES:
Resolution of symptoms and interferon gamma activity at 2 and 6 months | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Sushil Kr Kabra, MD, Principal Investigator — All India Institute of Medical Sciences
Locations (1):
- Department of Pediatrics, All India Institute of Medical Sciences, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lodha R, Mukherjee A, Singh V, Singh S, Friis H, Faurholt-Jepsen D, Bhatnagar S, Saini S, Kabra SK, Grewal HM; Delhi Pediatric TB Study Group. Effect of micronutrient supplementation on treatment outcomes in children with intrathoracic tuberculosis: a randomized controlled trial. Am J Clin Nutr. 2014 Nov;100(5):1287-97. doi: 10.3945/ajcn.113.082255. Epub 2014 Sep 10. PMID 25332327